CLINICAL TRIAL: NCT01598350
Title: Using Anthropometric Measurements to Predict Orthotic Influence on Gait Parameters in Children With Down Syndrome
Brief Title: Gait in Children With Down Syndrome While Wearing Orthoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puget Sound (Other)
Responsible Party: Principal Investigator, Julia Looper, Assistant Professor, University of Puget Sound
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0910-003
Record Dates: First submitted 2010-01-20; First posted 2012-05-15 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-11

CONDITIONS: Down Syndrome
Keywords: Gait; Orthoses; Down syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orthotic (Experimental): Orthotic Use
  Interventions: Device: Supramalleolar Orthoses (Cascade)

INTERVENTIONS:
Device: Supramalleolar Orthoses (Cascade) — Walk wearing supramalleolar orthoses - three trial
  Other Names: Cascade - leap frog

SUMMARY:
On average, Down syndrome (DS) occurs once in every 700 live births and results in life-long disability and increased risk for comorbidities.1 Individuals with DS are also susceptible to secondary physical impairments and limitations as a result of complications associated with joint hypermobility, hypotonicity, and increased ligamentous laxity. Secondary impairments such as pes planus (flat feet), weakened muscles, bony abnormalities and arthritis may lead to painful joints and feet. Additionally, children with DS often manifest deviations in gait as a result of physical limitations imposed by orthopedic and muscular deficiencies that may lead to decreased postural stability. These secondary losses in function, which exacerbate disabilities, may be preventable with the use of appropriate early interventions aimed at correcting abnormal joint alignment. Research exploring effective physical therapy interventions for adults and children with DS is currently very limited. However, the use of orthotic devices to support lax ligaments and hypotonic muscles, which are common manifestations of DS, is one accepted method of intervention for children within this population. Orthoses are variable in structure and the degree of support provided to the foot and ankle also differ between foot orthoses (FOs) and supramalleolar orthoses (SMOs). Previous studies have supported the effectiveness of orthoses on improving ankle and foot alignment, as well as gait parameters. However, disagreement currently exists concerning which type of orthotic device is most beneficial for the population of children with DS. Children with DS express variable degrees of joint laxity and hypotonicity, as well as differences in the severity of specific alignment abnormalities such as excessive pronation or calcaneal eversion.6 Current literature is insufficient for explaining differences in the benefits provided by FOs and SMOs and the specific indications for their use in children with DS is unclear.

Study Aims This study will demonstrate the differences in structural outcomes provided by FOs and SMOs and develop specific criterion for matching individuals of differing orthopedic impairments with the most beneficial orthotic device.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the differences in functional outcomes provided by supramalleolar orthoses and foot orthoses, as well as develop specific criterion for matching individuals with Down syndrome (DS) of differing orthopedic impairments with the most beneficial orthotic device.

Participants must be able to walk independently or with an assistive device, such as a walker, for 50 feet at one time, and have at least six months of walking experience. Participants must also be able to follow simple verbal instructions. Both males and females will be included in this study, and children of any race may participate as long as they meet the inclusion criteria and are between three and ten years of age at the time of data collection. Exclusion criteria include a history of uncorrected visual and inner ear impairments, and lower extremity orthopedic surgical corrections.

There are no costs associated with participation in this study, and subjects will not be paid for their participation.

Participants in this study will be fitted for the appropriate size orthoses either by physical therapists in the participants' school district, or by one of the researchers prior to data collection. The correct fitting orthotic will be sized using the sizing guides provided by Cascade. These are footplates of various sizes that provide the length of the child's foot in inches and the orthosis width that will fit the child. Measurements of height, weight, leg length, medial longitudinal arch height, tibial torsion, and calcaneal eversion will be taken for each subject. Weight will be measured in kilograms using a scale, while height, leg length, and medial longitudinal arch height will be measured using a metric tape measure. Tibial torsion will be measured with the participant lying in prone (on their stomach) on the plinth with one knee flexed to 90 degrees. The angle of tibial torsion is formed by a line perpendicular to the line between the medial and lateral malleoli of the ankle, and a line parallel to the femur. This angle will be measured using a goniometer, which is an instrument used to measure joint angles and range of motion, and this angle will be measured once on each side. Finally, while standing, calcaneal eversion will be measured by determining the angle between neutral calcaneal alignment and resting stance. Neutral calcaneal alignment is found by palpating the position of the talus, so that the talus bone is felt equally on both sides of the foot. Once neutral alignment has been determined a line will be drawn with washable marker between the posterior talus and midline of the calf. The participant will then be asked to stand in their normal position and a goniometer will be used to measure the angle between the neutral alignment and the resting alignment of the ankle.

In addition to these measurements, a hypermobility screen will be performed in which mobility of fingers, wrists, elbows, knees, and the spine will be scored. The screen is scored using a point system in which one point is given for the ability to perform each of the tasks in the screen. These tasks include the ability to actively extend the little fingers 90 degrees at the metacarpophalangeal joints, passively touch the thumbs to the volar surface of the forearms, extend the wrists more than 90 degrees, extend elbows and knees more than 10 degrees, and the ability to bend the spine to reach the floor with palms flat on the ground. Gait of each participant will be assessed in conditions of shoes only, with foot orthoses, and with supramalleolar orthoses. This order will be determined by selecting a condition at random from a hat, such that the first condition chosen will be performed and assessed first.

Gait parameters including step length, step width, walking speed, percentage of time spent in single leg support, and variability in gait will be measured using a GAITRite mat. The GAITRite measurement system includes an electronic walkway which contains sensor pads, and is similar to a roll-out carpet. The GAITRite mat is then linked to a computer, which collects information about gait as the participant walks across the mat. The GAITRite mat, which is 20 feet long, will be set-up as one segment of a circular track so that total walking distance of the loop will be 50 feet. Participants will be given an accommodation period of ten minutes for both types of orthoses prior to gait assessment in which they will be instructed to walk around the room and over the GAITRite mat in order to get comfortable wearing the orthoses and walking along the track. Once the accommodation period is complete for one orthosis, participants will walk around the track three times. This procedure of accommodation and data collection will be repeated for each condition. Participants will be given verbal encouragement by the researchers as they walk the track as a means of motivation. Rest periods will be given to participants when requested, or when behavioral cues displaying discomfort, pain, or frustration occur. Data collection will be stopped altogether at the participant's request or if behavioral cues of discomfort persist. Trials involving both supramalleolar and foot orthoses are hypothesized to increase step length, walking speed, and time spent in single leg support from control trials in the shoes only condition. Both orthoses are also expected to decrease step width, and variability in gait parameters. Supramalleolar orthoses, which provide above-ankle support, are expected to improve gait parameters to a greater magnitude than foot orthoses for participants who score higher on the hypermobility screen and have greater tibial torsion and ankle eversion than their cohorts. Conversely, foot orthoses are expected to provide greater improvement in gait parameters than supramalleolar orthoses for participants who score lower on the hypermobility screen and have less tibial torsion and ankle eversion than their cohorts due to the need for less external foot and ankle support. An increase in step length, walking speed, time spent in single leg support, and a decrease in step width and variability in gait will indicate a positive result of orthoses use.

Students of physical therapy from the University of Puget Sound Physical Therapy Program will perform all measurements, with the exception of orthotic size in some cases. One researcher will perform all anthropometric measurements and the hypermobility screen on the participants. A second researcher will operate the GAITRite mat, while the third researcher will guide and instruct the participants along the GAITRite mat course.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to walk independently or with an assistive device, for 50 feet at one time, and have at least six months of walking experience. Participants must also be able to follow simple verbal instructions.

Exclusion Criteria:

* Exclusion criteria include a history of uncorrected visual and inner ear impairments, and lower extremity orthopedic surgical corrections.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puget Sound, Tacoma, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from local elementary schools from November 2009 until January 2009
Groups:
- Orthotic: Orthotic Use
  Supramalleolar Orthoses (Cascade) : Walk wearing supramalleolar orthoses - three trial
Period: Overall Study
Arm/Group | Orthotic
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Orthotic
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 4.5 (.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Step Width
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Orthotic
Number analyzed (Participants) | 6
cm | 10.4 (2.8)

ADVERSE EVENTS:
Arm/Group | Orthotic
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
small number of subject recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes